CLINICAL TRIAL: NCT06005077
Title: Evaluation of the Effect of Perineal Massage and Warm Application on Perineal Trauma, Pain and Birth Comfort in Labor
Brief Title: Perineal Massage and Warm Application in Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Gamze Acavut, Asst. Prof, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/13
Record Dates: First submitted 2023-01-30; First posted 2023-08-22 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Perineal Injury; Pain; Labor
Keywords: Labor; Perineal massage; Perineal warm compress; Perineal Trauma
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The patients and principle investigator knew which group they were assigned to. Only the outcome assessor didn't know which patient was assigned to which group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): After the hospitalization procedures were completed, the pregnant women in the control group were informed and their written consents were obtained. No intervention was performed on these pregnant women other than routine hospital practices. Data collection forms were applied.
- Perineal Massage (Experimental): While the pregnant woman was in the lithotomy position, massage was applied with two fingers and rhythmic U-shaped movements starting from the side walls 3-4 cm inside the vagina and towards the rectum. This implementation was done for 10 minutes in three stages according to cervical dilatation. It was applied when the cervical dilatation was 3-4 cm, 5-7 cm, and 8-10 cm.
  Interventions: Other: Perineal Massage Group
- Perineal Warm Compress Application (Experimental): Sterile compresses kept in hot water of 40 C were placed on the perineum. Compresses that cooled down and became dirty were changed every 5-8 minutes. This implementation was done for 30 minutes in three stages according to cervical dilatation. It was applied when the cervical dilatation was 3-4 cm, 5-7 cm, and 8-10 cm.
  Interventions: Other: Perineal Warm Compress Application Group
- Perineal Massage and Perineal Warm Compress Application (Experimental): When the cervical dilatation was 3-4 cm, 30 minutes of warm compress and 10 minutes of perineal massage were performed. These two methods were applied when the cervical dilatation was 5-7 cm and 8-10 cm as well.
  Interventions: Other: Perineal Massage Group; Other: Perineal Massage and Perineal Warm Compress Application Group

INTERVENTIONS:
Other: Perineal Massage Group — While the pregnant woman was in the lithotomy position, massage was applied with two fingers and rhythmic U-shaped movements starting from the side walls 3-4 cm inside the vagina and towards the rectum. This implementation was done for 10 minutes in three stages according to cervical dilatation. It was applied when the cervical dilatation was 3-4 cm, 5-7 cm, and 8-10 cm.
  Arms: Perineal Massage; Perineal Massage and Perineal Warm Compress Application
Other: Perineal Warm Compress Application Group — Sterile compresses kept in hot water of 40 C were placed on the perineum. Compresses that cooled down and became dirty were changed every 5-8 minutes. This implementation was done for 30 minutes in three stages according to cervical dilatation. It was applied when the cervical dilatation was 3-4 cm, 5-7 cm, and 8-10 cm.
  Arms: Perineal Warm Compress Application
Other: Perineal Massage and Perineal Warm Compress Application Group — When the cervical dilatation was 3-4 cm, 30 minutes of warm compress and 10 minutes of perineal massage were performed. These two methods were applied when the cervical dilatation was 5-7 cm and 8-10 cm as well .
  Arms: Perineal Massage and Perineal Warm Compress Application

SUMMARY:
The aim of this study is to determine the effect of perineal massage and warm compress application at first and second stage of labor on perineal trauma, pain and delivery comfort.

DETAILED DESCRIPTION:
Perineal trauma is the damage caused by rupture, laceration or episiotomy during birth. Birth-related perineal trauma can lead to many short and long-term physical and psychological morbidities that affect the woman's life. Problems such as pain, bleeding and delay in the attachment of mother and newborn appear in the early postpartum period. In the following period problems such as prolapse, incontinence, sexual dysfunction and anxiety may be experienced.

This randomised controlled study was executed at a research hospital between May 2018 - September 2019. The sample of study is made consisted of three intervention groups and a control group of total 120 pregnant women by randomisation method. Perineal massage, perineal warm compress application, perineal massage and warm compress was done to the intervention groups respectively. Nothing was done to the control group. Perineal massage was given for 10 minutes, warm compress application was done 30 minutes three times when cervical dilatation 3-4 cm, 5-7 cm and 8-10 cm respectively. The data was collected by using Socio-Demographic and Obstetric Data Collection Form, First and Second Stage of Labor Stage Data Collection Form, Childbirth Comfort Scale, Newborn Data Collection Form, Perineal Trauma and Bleeding Monitorisation/ Measurement Form, Visual Analogue Scale, Birth Satisfaction Scale and Perineal Massage and Perineal Warm Compress Application Satisfaction Evaluation Form. When evaluating the data; number, percentage, mean, standard deviation, median, ANOVA Test, Tukey Test, Kruskal Wallis Test, Paired Sample T Test, Friedman Test, Ki-Square Test and Fisher's Exact was used.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous
* 38"week of pregnancy
* Singleton pregnancy
* Cervical dilatation 3"cm
* Cephalic presentation

Exclusion Criteria:

* Chronic disease
* Presence of fetal macrosomia
* Presence of uterin surgery
* Presence of fetal anomaly

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only women who were going to give birth were included in the study.
Enrollment: 120 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Socio-Demographic and Obstetric Data Collection Form | Baseline
  The Socio-Demographic and Obstetric Data Form was used to determine the socio-demographic and obstetric characteristics of the participants. This form, created by the investigators, includes 15 questions on age, height, weight, education level, and gestational week of the pregnant women, the way pregnancy occured, and the health problems experienced during pregnancy.
First and Second Stage of Labor Stage Data Collection Form | During procedure
  The First and Second Stage of Labor Data Form and the Newborn Data Form were used to note down the applications performed on the pregnant woman during the first and second stages of labor and on the newborn after delivery. The form created by the investigators following the review of the literature consists of three parts. In the first part, there are questions regarding the applications such as dilatation, wiping, drugs used in the first stage, amniotomy, and bladder catheterization performed when the pregnant woman is admitted into the delivery room. In the second part, there are questions on the application of local anesthesia in the second stage of labor, protection of the perineum, and the type of pushing. The third part consists of questions regarding the height, weight and APGAR measurement of the newborn. This form includes 33 questions in total.
Childbirth Comfort Scale | During the procedure
  The Childbirth Comfort Scale (CCS) is used to determine the comfort level at birth. This scale is a 5-point Likert type scale and consists of 14 items. Each item is rated between 1-5 (1: Strongly disagree, 2: Mostly disagree, 3: Partially agree, 4: Mostly agree, 5: Completely agree). The scale has a four-factor structure: physical, psychospiritual, social and environmental.
Birth Satisfaction Scale | In the first 1 hour after birth
  The Birth Satisfaction Scale (BSS) is used to evaluate birth satisfaction. This scale is a 5-point Likert-type scale and consists of 30 items. The three main themes of the scale are quality of care, personal characteristics of the women, and stress experienced during childbirth. A minimum of 30 and a maximum of 150 points can be obtained from the scale. Higher scores indicate higher levels of satisfaction.
Perineal Trauma and Bleeding Monitorisation/Measurement Form | In the first 1 hour after birth
  The Perineal Trauma, Postpartum Bleeding and Episiotomy Length Evaluation Form was used to record data on perineal trauma and amount of bleeding. The form, created by theinvestigators, consists of 13 questions evaluating conditions such as episiotomy, type of perineal trauma, location and degree of trauma, and postpartum bleeding.
Visual Analogue Scale | During procedure
  The Visual Analog Scale (VAS) is a one-dimensional measurement tool used to show perceived pain and its severity. One end of the scale indicates "painlessness (0)" and the other end indicates "the most severe pain possible (10)" .
Birth Satisfaction Scale | In the first 1 hour after birth
  The Newborn Characteristics Data Collection Form consists of 7 questions including the newborn's height, weight and APGAR assessment.
Perineal Massage and Perineal Warm Compress Application Satisfaction Evaluation Form | In the first 1 hour after birth
  This form was used to record the phases, periods and durations of perineal massage and perineal heat application, as well as to evaluate the satisfaction with the application. A visual scale graded from 0 to 10 was used in the satisfaction evaluation. It was rated as "0" not at all satisfied, "10" very satisfied.In addition, the participants were asked whether the application was beneficial, whether participants would prefer it when they gave birth again, and whether they would recommend it to others. It was created by the researcher and expert approval was obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Acavut, Principal Investigator — Ankara Medipol University
Locations (1):
- Gamze Acavut, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ducarme G, Pizzoferrato AC, de Tayrac R, Schantz C, Thubert T, Le Ray C, Riethmuller D, Verspyck E, Gachon B, Pierre F, Artzner F, Jacquetin B, Fritel X. Perineal prevention and protection in obstetrics: CNGOF clinical practice guidelines. J Gynecol Obstet Hum Reprod. 2019 Sep;48(7):455-460. doi: 10.1016/j.jogoh.2018.12.002. Epub 2018 Dec 12. PMID 30553051
- [Background] Fukami T, Koga H, Goto M, Ando M, Matsuoka S, Tohyama A, Yamamoto H, Nakamura S, Koyanagi T, To Y, Kondo H, Eguchi F, Tsujioka H. Incidence and risk factors for postpartum hemorrhage among transvaginal deliveries at a tertiary perinatal medical facility in Japan. PLoS One. 2019 Jan 9;14(1):e0208873. doi: 10.1371/journal.pone.0208873. eCollection 2019. PMID 30625154
- [Background] Barasinski C, Debost-Legrand A, Lemery D, Vendittelli F. Practices during the active second stage of labor: A survey of French midwives. Midwifery. 2018 May;60:48-55. doi: 10.1016/j.midw.2018.02.001. Epub 2018 Feb 8. PMID 29494852
- [Background] Difranco JT, Romano AM, Keen R. Care practice #5: spontaneous pushing in upright or gravity-neutral positions. J Perinat Educ. 2007 Summer;16(3):35-8. doi: 10.1624/105812407X217138. PMID 18566649
- [Derived] Acavut G, Guvenc G, Karasahin KE. The Effectiveness of Massage and Warm Compresses on Perineal Trauma, Hemorrhage, Length of Episiotomy and Pain: A Randomized Controlled Trial. Z Geburtshilfe Neonatol. 2025 Nov 19. doi: 10.1055/a-2730-1313. Online ahead of print. PMID 41260484